CLINICAL TRIAL: NCT06123455
Title: A Prospective, Randomized Controlled Clinical Study of The Efficacy and Safety of Taurine Combined With Sintilimab and Chemotherapy Versus Sintilimab Combined With Chemotherapy for Treatment of Advanced Gastric Cancer
Brief Title: Clinical Study of Taurine Combined With Sintilimab and Chemotherapy for Treatment of Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K202309-06
Record Dates: First submitted 2023-09-20; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Taurine; sintilimab; XELOX; Folfox protocol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taurine + Sintilimab + investigator's choice chemotherapy (Experimental): Taurine + Sintilimab + XELOX or Taurine + Sintilimab + SOX or Taurine + Sintilimab + FOLFOX
  Interventions: Dietary Supplement: Taurine; Biological: Sintilimab; Drug: XELOX regimen; Drug: SOX regimen; Drug: FOLFOX regimen
- Sintilimab + investigator's choice chemotherapy (Active Comparator): Sintilimab + XELOX or Sintilimab + SOX or Sintilimab + FOLFOX
  Interventions: Biological: Sintilimab; Drug: XELOX regimen; Drug: SOX regimen; Drug: FOLFOX regimen

INTERVENTIONS:
Dietary Supplement: Taurine — Taurine supplementation in capsules of 1.0 gram of taurine powder. Dosage: 2.0 gram/day. Frequency: 2 time/day.
  Arms: Taurine + Sintilimab + investigator's choice chemotherapy
Biological: Sintilimab — Sintilimab
Drug: XELOX regimen — Oxaliplatin + capecitabine
Drug: SOX regimen — Oxaliplatin + S-1 (tegafur/gimeracil/oteracil potassium)
Drug: FOLFOX regimen — Oxaliplatin + leucovorin + fluorouracil

SUMMARY:
This project aims to evaluate the efficacy and safety of oral taurine supplementation combined with PD-1 inhibitor (sintilimab) and chemotherapy in inducing systemic CD8+ T cell responses and achieving improved gastric cancer patient outcomes than with sintilimab and chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older, no gender limitation;
2. Pathologically confirmed gastric cancer or adenocarcinoma of the gastroesophageal junction, local lesions cannot be radically resected or metastatic gastric cancer;
3. Expected survival of ≥ 3 months;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
5. At least one measurable lesion outside the stomach (RECIST 1.1);
6. Patients informed about the purpose and course of the study and provided a written consent to participate.

Exclusion Criteria:

1. Use of taurine agent within 1 month prior to randomization on this study;
2. Patients received prior systemic therapy for gastric cancer;
3. Patients with operable gastric cancer;
4. Patients with positive HER-2 and willing to receive herceptin treatment;
5. Patients with gastrointestinal obstruction or active bleeding in the gastrointestinal tract, as well as perforation and dysphagia;
6. Patients with active autoimmune disease that has required systemic treatment in past 2 years;
7. Patients diagnosed as immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy;
8. Patients with severe heart, lung, liver, kidney, endocrine, hematopoietic system or psychiatric diseases were considered not suitable for the study group;
9. Patients with other medical conditions that interfere with the trial and are deemed unsuitable for inclusion in the trial by the investigator;
10. Other conditions that the investigator thinks are not suitable to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 24 months
  PFS was defined as the time from randomization to the first documented disease progression (PD) per RECIST 1.1 based on independent radiology review or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 24 months
  OS was defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months
  ORR is defined as the proportion of subjects with complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.
Safety profile | Up to 24 months
  Number of study subjects experiencing adverse events (AEs), dose-limiting toxicities, and serious adverse events (SAEs). Safety profile will be assessed through laboratory evaluations, vital signs, and physical examinations.

OTHER OUTCOMES:
Changes in CD8+ T cell death and function | Up to 24 months
  Changes in number, apoptosis rate, effector (TNF-α, IFN-γ, etc.) production and immune checkpoint molecule (PD-1, CTLA-4, etc.) expression of CD8+ T cells in peripheral venous blood assessed via flow cytometry.
Changes in CD8+ T cell infiltration in tumor tissue | Up to 24 months
  Changes in number, effector (TNF-α, IFN-γ, etc.) production and immune checkpoint molecule (PD-1, CTLA-4, etc.) expression of tumor-infiltrating CD8+ T cells in gastric cancer endoscopic biopsy material assessed via immunohistochemistry.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Wang, MD, PhD, Study Director — Tang-Du Hospital; Xiaodi Zhao, MD, PhD, Principal Investigator — Xi-Jing Hospital; Yuanyuan Lu, MD, PhD, Principal Investigator — Xi-Jing Hospital
Locations (1):
- Tang-Du Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No